CLINICAL TRIAL: NCT05590546
Title: Concomitantly Higher Resting Arterial Blood Pressure and Transduction of Sympathetic Neural Activity in Human Obesity Without Hypertension
Brief Title: Sympathetic Transduction in Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Seth Holwerda PhD, Assistant Professor, University of Kansas Medical Center
Other Study IDs: TRANSDUCTION_IN_OBESITY
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese: No intervention, only performing cross-sectional analysis of pooled data collected in previous studies
  Interventions: Other: No intervention
- Control: No intervention, only performing cross-sectional analysis of pooled data collected in previous studies
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, only performing cross-sectional analysis of pooled data collected in previous studies

SUMMARY:
Central (abdominal) obesity is associated with elevated adrenergic activity and arterial blood pressure (BP). Therefore, we tested the hypothesis that transduction of spontaneous muscle sympathetic nerve activity (MSNA) to BP, i.e., sympathetic transduction, is augmented in abdominal obesity (increased waist circumference) and positively related to prevailing BP.

DETAILED DESCRIPTION:
The prevalence of obesity has increased to over 42% of adults in the United States. Obesity, particularly elevations in central adiposity, is associated with the development of hypertension, which is a prominent cause of cardiovascular diseases (CVD), such as stroke, myocardial infarction, heart failure, and chronic kidney disease. Pathophysiology of obesity hypertension includes several different categories of mechanisms, such as sympathetic activation, inflammation, and renal dysfunction. However, the relative importance and contribution of these mechanisms to the initiation of obesity hypertension remains uncertain.

Obesity is characterized by elevated peripheral vascular tone. Specifically, larger decreases in arterial blood pressure (BP) were observed following ganglionic blockade (trimethaphan) in obese individuals compared with non-obese controls, suggesting greater autonomic support of BP in obesity. Similarly, 4 weeks of combined α- and β-adrenergic receptor blockade produced larger reductions in BP in obese participants with hypertension compared with non-obese control with hypertension. These data are consistent with the large body of evidence suggesting that obesity elevates muscle sympathetic nerve activity (MSNA). However, MSNA may not be elevated in obesity if development of hypertension is absent. Therefore, the extent to which MSNA contributes to the initial development of BP dysregulation in obese men and women without hypertension remains unclear.

Obesity-related increases in vascular tone may be, in part, a result of increased vascular responsiveness to MSNA. In fact, elevated vascular responsiveness to MSNA has been reported in obesity-related conditions such as type 2 diabetes. However, only one study has directly examined sympathetic vascular tone in obese subjects without hypertension, reporting similar passive increases in forearm blood flow following α-adrenergic receptor blockade when compared to age- and sex-matched non-obese participants. These data suggest that obesity alone does not alter passive dilation of the forearm resulting from α-adrenergic receptor blockade. However, an extrapolation to systemic BP regulation in obesity from an examination of forearm dilation is challenging for several reasons. First, passive dilation following α-adrenergic receptor blockade may not reflect the blood flow response to α-adrenergic receptor activation, i.e., endogenous sympathetic activation. Second, in normal adults, vascular responsiveness to sympathetic innervation is heterogenous across vascular regions. For example, the lower limbs exhibit greater vascular sensitivity to sympathetic stimulation compared with the forearm vasculature as a result of greater α-adrenergic receptor density and/or sensitivity in the lower limbs. Third, obese individuals exhibit regional differences in endogenous norepinephrine kinetics compared with non-obese individuals. Thus, although regional sympathetic vascular tone has been assessed in obesity, there are limited data available regarding potential alterations in systemic BP responsiveness to endogenous activation of adrenergic receptors in this population who are highly prone to development of hypertension.

Therefore, a technique that quantifies the systemic pressor response to spontaneous bursts of MSNA with high temporal resolution (i.e., sympathetic transduction) is used. It is hypothesized that sympathetic transduction would be augmented in young/middle-aged men and women with abdominal obesity (increased waist circumference) compared with age- and sex-matched non-obese controls. It is further hypothesized that augmented sympathetic transduction in obesity would be positively related to higher prevailing BP.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers
* free of metabolic or neurological disease
* waist circumference > 102 cm for men and > 88 cm for women or waist circumference was < 94 cm for men and < 80 cm for women.

Exclusion Criteria:

* Use of anti-hypertensive medications
* history of diabetes
* history of smoking within 3 months prior to study participation
* hypertension determined by 24-hour ambulatory average BP (<130/80 mmHg).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Otherwise healthy
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Sympathetic transduction | 15 min
  signal averaging was performed in which bursts of MSNA act as a trigger and beat-to-beat BP was tracked for 15 subsequent cardiac cycles thereafter.

IPD SHARING:
Plan to Share IPD: Undecided